CLINICAL TRIAL: NCT00643045
Title: A Phase III, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of a Low (50 100 mg/Day) and High (150 200 mg/Day) Dose Range of Safinamide as Add-On Therapy in Patients With Early Idiopathic Parkinson's Disease Treated With a Stable Dose of a Single Dopamine Agonist
Brief Title: Safinamide as Add-On Therapy in Patients With Early Idiopathic Parkinson's Disease Treated With a Stable Dose of a Single Dopamine Agonist
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Dr Stefano Rossetti, Newron Pharmaceuticals S.p.A.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NW 1015/015/III/2003
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Low dose (50-100mg/day)
  Interventions: Drug: Safinamide
- 2 (Experimental): High dose (150-200 mg/day)
  Interventions: Drug: Safinamide
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Safinamide
  Arms: 1
Drug: Safinamide
  Arms: 2
Drug: Placebo
  Arms: 3

SUMMARY:
To evaluate the safety and efficacy of two dose ranges of safinamide (High Dose: 150 to 200 mg/day and Low Dose: 50 to 100 mg/day) orally, as compared to Placebo, as add-on therapy in patients with early idiopathic Parkinson's disease who are currently receiving a stable dose of a single dopamine agonist. It is hypothesized that, over a 24-week period, add-on treatment with safinamide will result in greater improvement of motor symptoms in these patients, compared to treatment with a dopamine agonist alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of idiopathic Parkinson's disease of less than 5 years duration, and a Hoehn and Yahr Stage of I to III,
* who were receiving treatment with a single dopamine agonist at a stable dose for at least 4 weeks prior to Visit 1 (Screening).

Exclusion Criteria:

* Patients with medical conditions and/or taking concomitant medications that would have put them at risk, interfered with the study evaluations, or made them unable to complete the requirements of the study;
* patients with a diagnosis or recent history of substance abuse,
* a history of psychosis,
* who were depressed,
* had evidence of dementia or cognitive dysfunction,
* or who were experiencing end of dose wearing-off;
* female patients of childbearing potential;
* patients who have previously received safinamide.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 269 (Actual)
Dates: Start 2004-12; Primary Completion 2006-01 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
UPDRS Section III (Motor Examination [ME]) total score at Baseline, each post-baseline visit and Endpoint (Visit 8 [Week 24]). | 24 weeks

SECONDARY OUTCOMES:
UPDRS Section III (ME) item (& total) scores.CGI Change from Baseline score.UPDRS Section II (ADL) item (& total) scores.CGI Severity of Illness score. H&Y Staging.All above at each visit and Endpoint (LOCF). Cogtest PD battery score each visit | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Merello, MD, Principal Investigator — Instituto FLENI, Buenos Aires; Rolando Giannaula, MD, Principal Investigator — Hospital Español - Servicio de Neurologia, Buenos Aires; Federico Micheli, MD, Principal Investigator — Hospital de Clinicas, Servicio de Movimientos, Buenos Aires; Marcelo Miranda, MD, Principal Investigator — Liga Chilena Contra el Mal De Parkinson, Santiago, Chile; David Saez, MD, Principal Investigator — Hospital Barros Luco Trudeau, Servicio de Neurologia, Santiago, Chile; Roque Villagra, MD, Principal Investigator — Hospital Salvador-Neurologia, Santiago, Chile; Yuri Takeuchi, MD, Principal Investigator — Fundaciόn Valle de Lili Direcciόn Médica, Cali-Valle, Colombia; Mauricio Acevedo, MD, Principal Investigator — Hospital Militar, Departamento de Neurología, Bogotà-D.C, Colombia; Pablo Lorenzana, MD, Principal Investigator — Consultorio, Bogotà-D.C, Colombia; Madhuri Behari, MD, Principal Investigator — Department of Neurology, All India Institute of Medical Science (AIIMS), New Delhi, India; Mohit Bhatt, MD, Principal Investigator — Movement Disorder Clinic, Jaslok Hospital, Mumbai, India; Rupam Borgohain, MD, Principal Investigator — Nizam's Institute of Medical Sciences (NIMS), Hyderabad, India; Arunkumar Shah, MD, Principal Investigator — B.Y.L. Nair Hospital & T.N. Medical College, Mumbai, India; Ajit Roy, MD, Principal Investigator — St John's Medical College & Hospital, Bangalore, India; Uday Babu Rao Muthane, MD, Principal Investigator — National Institute of Mental Health and Neuro Sciences, Bangalore, India; Fabrizio Stocchi, MD, Principal Investigator — IRCCS Neuromed Via Atinense 18 Pozzilli (IS), Italy; Leonardo Scarzelia, MD, Principal Investigator — Ospedale Evangelico Valdese, Torino, Italy; Gianpietro Nodera, MD, Principal Investigator — Dipartimento di Neurologia Casa di Cura "Villa Margherita", Vicenza, Italy; Pezzoli, MD, Principal Investigator — Isituti Clinici di Perfezionamento Centro Parkison, Milano, Italy; Leontino Battistin, MD, Principal Investigator — Dipartimento di Neuroscienze, Padova, Italy; Marco Onofri, MD, Principal Investigator — Divisione di Neurologia, Ospedale civile di Pescara, Italy; Paolo Lamberti, MD, Principal Investigator — Clinica Neurologica I Policinico di Bari, Italy; Alessandra Monge, MD, Principal Investigator — Osp. S. Giovanni Battista, Roma, Italy; Paolo Barone, Prof, MD, Principal Investigator — Dipartimento di Scienze Neurologiche, Universita di Napoli Federico II, Naples, Italy; Giovanni Abruzzese, MD, Principal Investigator — Dipartimento di Neuroscienze DINOG, Universita degli Studi di Genova, Italy; Roberto Marconi, MD, Principal Investigator — Ospedale della Misericordia, Grosseto, Italy; Kulisevsky, MD, Principal Investigator — Serv. Neurologia, Barcelona, Spain; Lopez Lozano, MD, Principal Investigator — H. Puerta de Hierro, Serv. Neurologia, Madrid, Spain; Antonio Vacquez, MD, Principal Investigator — H. Clinico San Carlos, Ser. Neurologia, Spain; Schapira, Prof, MD, Principal Investigator — Department of Neurology, Royal Free Hospital, UK; Chaudhuri, MD, Principal Investigator — Day Hospital, Care of the Elderly, Lewisham University Hospital, London, UK; Barker, MD, Principal Investigator — Cambridge Centre for Brain Repair, Cambridge, UK